CLINICAL TRIAL: NCT03544346
Title: An Investigation Into the Long-term Brain Health of Retired Professional Rugby Players, With a History of Concussion/Head Impact Exposure
Brief Title: Long-term Brain Health of Retired Professional Rugby Players, With a History of Concussion/Head Impact Exposure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Joice Cunningham, Ms Joice Cunningham (Phd Candidate), University of Dublin, Trinity College
Other Study IDs: JCunningham
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Brain Health Retired Elite Athletes
Keywords: brain health, professional athlete, retired, neuropsychological assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retired professional rugby players: Rugby Players will Provide detailed demographic information Provide detailed overall health information Questionnaires Provide information on athlete's playing career; age of debut, career duration, number of seasons participated in. Provide information on concussion history. Be given a general health screen including- heart rate, blood pressure, body composition and height weight ratio.
  Perform a battery of neuropsychological tests (Sound-induced flash illusion and CANTAB, NART) Provide a sample of blood.
  Interventions: Other: Exploratory brain and general health assessment
- Retired professional rowers: Rowers will Provide detailed demographic information Provide detailed overall health information Questionnaires Provide information on athlete's playing career; age of debut, career duration, number of seasons participated in. Provide information on concussion history. Be given a general health screen including- heart rate, blood pressure, body composition and height weight ratio.
  Perform a battery of neuropsychological tests (Sound-induced flash illusion and CANTAB, NART) Provide a sample of blood.
  Interventions: Other: Exploratory brain and general health assessment

INTERVENTIONS:
Other: Exploratory brain and general health assessment — Exploratory brain and general health assessment

SUMMARY:
There has been significant recent interest on the issue of brain health in athletes. Participation in sports is generally viewed as extremely positive. Consistent evidence supports associations among exercise, cognitive vitality, neural functioning and decreased risk of cognitive decline. However, In the last decade, a dramatic shift in both public and scientific perception around the long-term consequences of concussion is evident. Rugby is a popular full-contact sport played throughout the world at varying levels of competition, including professional level. The game exposes players to inherent risk of injury including repetitive head impacts, due to the high number of collisions and tackles involved. Perhaps not surprisingly, given the physical nature of the sport, rugby has one of the highest rates of concussion of all full-contact sports. Evidence from a recent meta-anaysis found the incidence of concussion to be 4.73 per 1000 player match hours. Given the high incidence of concussion that has been reported in the literature to date, the issue of concussion and repeated head impact exposure is of particular concern in rugby.

Comprehensive investigation of cognition in living retired sports persons with previous exposure to repetitive head impact is noticeably lacking in the literature to date. Findings are inconsistent and investigations are shrouded by consistent methodological biases and flaws, reducing the overall quality of the studies. Relatively little research has been conducted on the long-term effects of repetitive mild TBI or sports concussion on the retired athlete's brain health with ageing. The potential long-term consequences are poorly understood and warrant more research. This study aims to investigate the brain health of retired rugby players in comparison to retired rowers who have achieved the same levels of exercise, without exposure to SRCs

DETAILED DESCRIPTION:
The primary aim of this study is to investigate brain health and wellness of retired professional Irish rugby players in comparison to retired professional Irish rowers.

Objectives:

The objectives will be to:

Obtain detailed demographic and overall health information from the retired rugby players and retired rowers.

Use a battery of cognitive function tests to assess the cognitive health of the retired rugby players and retired rowers.

Obtain blood samples from the retired rugby players and retired rowers in order to test for biomarkers indicative of neurodegenerative disease.

Investigate rugby player's self-report history of sports-related concussion (number and nature of concussions) during their career. Player's self-report will be correlated where possible with established individual player medical data.

ELIGIBILITY:
Inclusion Criteria:

- Male A retired professional rugby player (no age limit), who has played at least one season of professional rugby. A retired international rower (no age limit), who completed and trained full time for at least one season.

Athletes who have given informed consent and are willing to participate in the study.

Exclusion Criteria:

- You have a history of a non-sports related moderate to severe concussion or brain injury (eg a motor vehicle accident) You have had a concussion in the last year. You have had treatment of chemotherapy or radiotherapy in last 12 months. You have a bleeding disorder (will exclude you from blood sampling only).

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male
Study Population: Professional sport athletes with a career in elite rowing or rugby
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-18 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Brain Health Assessment | 1 hour
  Investigating cognitive functioning

SECONDARY OUTCOMES:
Concussion History Assessment | 20 minutes
  History of concussion/head impact exposure

IPD SHARING:
Plan to Share IPD: No